CLINICAL TRIAL: NCT01962181
Title: Identifying Characteristic Signature of Brain Activity of Electroencephalogram Records in Attention Deficit / Hyperactivity Disorder (ADHD) and Ritalin Treatment
Brief Title: Identifying Characteristic Signature of Attention Deficit / Hyperactivity Disorder (ADHD) and Ritalin Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RE0379-HMO-STILL
Record Dates: First submitted 2013-09-15; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-09

CONDITIONS: "Attention Deficit Hyperactivity Disorder"
Keywords: EEG Attention Deficit / Hyperactivity Disorder (ADHD) Ritalin machine learning
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ritalin (Active Comparator): Ritalin treatment at different doses
  Interventions: Drug: Ritalin
- Placebo (Placebo Comparator): Two meetings, one of which will be given a placebo and the other will be given a low dose of Ritalin, randomly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ritalin — Patients with ADHD and healthy subjects will be examined under Ritalin or placebo
  Arms: Ritalin
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this study we try to identify the signature of brain activity in the EEG of attention deficit disorder (ADHD) patients compared to healthy subjects under different doses of Ritalin (methylphenidate) treatment.

DETAILED DESCRIPTION:
In this study we try to identify the signature of brain activity in the EEG of attention deficit disorder (ADHD) patients compared to healthy subjects under different doses of Ritalin (methylphenidate) treatment. All subjects will undergo 1-4 EEG sessions. In each session we will use a different dose of Ritalin or placebo. A detailed neuropsychological tests will be done during the EEG recording. A powerful machine-learning techniques will be used in order to find a specific signature of ADHD and Ritalin treatment in the EEG recording.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, aged 18-50 years.
* Subjects aged 18-50 years diagnosed with ADHD and treated with Ritalin regularly (at least once a week).

Exclusion Criteria:

* Patients previously diagnosed as suffering from a brain disease except for ADHD.
* Patients after traumatic head injury.
* Patients who are unable to express their consent to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Resting oscillation activity and Event-related-Potentials in Attention Deficit / Hyperactivity Disorder (ADHD) and healthy subjects. | 2 years
  The primary outcome measure is the difference in the analysis of EEG recording (for example, resting oscillation activity and Event-related-Potentials) in Attention Deficit / Hyperactivity Disorder (ADHD) vs. healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Renana Eitan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel, Israel